CLINICAL TRIAL: NCT05226260
Title: Decreasing Antibiotic Duration for Skin and Soft Tissue Infections in Pediatric Primary Care Using Behavioral Economics Methods, A Cluster Randomized Trial
Brief Title: Decreasing Antibiotic Duration for Skin and Soft Tissue Infection Using Behavioral Economics in Primary Care
Acronym: SSTIBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joshua Watson, Principal Investigator, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00001964
Record Dates: First submitted 2021-11-03; First posted 2022-02-07 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cellulitis; Abscess; Drain Abscess; Impetigo; Skin Infection; Antibiotic Duration; Behavioral Economics
MeSH Terms: conditions — Cellulitis; Abscess; Impetigo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention clinics receiving fully functional Epic order panel with set default [short] duration by diagnosis: for cellulitis and drained abscess, 5 days. For impetigo and undrained abscess, 7 days.
  Interventions: Behavioral: Default Duration order Panel
- Control (No Intervention): Control clinics receiving basic Epic order panel with antibiotic doses by diagnosis but duration free text (must be entered manually by clinician prescriber).

INTERVENTIONS:
Behavioral: Default Duration order Panel — The SSTI order panel will present itself when a provider types in either a drug name or diagnosis (cellulitis, impetigo, etc). Clinicians in control clinics will have access to a basic order panel which will include diagnosis and corresponding antibiotic of choice. Clinicians in intervention clinics will have access to order panels with the following additional components: prepopulated order duration fields that default to the recommended treatment duration.
  Arms: Intervention

SUMMARY:
Study the efficacy of a package of behavioral economics strategies (versus an education-only control condition) in altering clinician behavior regarding antibiotic prescription duration for skin and soft tissue infection (SSTI).

DETAILED DESCRIPTION:
The investigators propose a prospective, cluster randomized trial of Epic order panels in the 14 Nationwide Children's Hospital (NCH) primary care clinics. Investigators have designed user-friendly Epic order panels from which providers may select guideline concordant antibiotics by simply typing in a diagnosis (cellulitis) or antibiotic name. These order panels are prepopulated with the default, short-course (guideline-concordant) antibiotic duration, saving clinicians several clicks within the electronic medical record (EMR). If a provider changes the prescribed duration from the one defaulted, a free text box will appear for them to write an acknowledgement reason (accountable justification). All 14 clinics will receive baseline education (control condition) about common infections and local and national guidelines for antibiotic choice and duration of treatment. Clinician prescribers will also be instructed about the presence of a basic order panel. The full functionality of the default [short/desired] duration order panel will only be released to intervention clinics. The order panels will be restricted in Epic to clinics randomized to the intervention. The investigators hypothesize that clinics with the intervention will have higher rates of short course antibiotics for SSTI versus control clinics.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis codes A46 (cellulitis), L03 (cellulitis and acute lymphangitis), J34 or L02 (abscess, furuncle), or L01 (impetigo) AND
* those who received a prescription for an enteral antibiotic
* patient's treated in Nationwide Children's Hospital primary care clinics

Exclusion Criteria:

* Patients less than 3 months of age
* Animal bite
* Human bite
* Foreign body
* Diagnosis of hidradenitis suppurativa
* Immunocompromising conditions (primary immune deficiency, chemotherapy, etc)
* burns

Ages: 3 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1634 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Rate of short antibiotics | 12 months
  Rates of long and short antibiotics will be analyzed on the clinic and provider level for both intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Kali Broussard, MD, Principal Investigator — Nationwide Children's Hospital; Joshua Watson, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital Primary Care Clinics, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Broussard KA, Chaparro JD, Erdem G, Abdel-Rasoul M, Stevens J, Watson JR. Default Antibiotic Order Durations for Skin and Soft Tissue Infections in Outpatient Pediatrics: A Cluster Randomized Trial. J Pediatric Infect Dis Soc. 2025 Jan 20;14(1):piae127. doi: 10.1093/jpids/piae127. PMID 39665614

DOCUMENTS (1):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT05226260/Prot_000.pdf